CLINICAL TRIAL: NCT00834912
Title: Study of Two Tramadol Contramid® OAD 300 mg Controlled-Release Tablets From Two Different Manufacturing Sites Following a 300 mg Dose in Healthy Subjects Under Fasting and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: MDT1-016
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-10-19 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Healthy Subjects
MeSH Terms: interventions — Tramadol

ARMS (3):
- 1: Tramadol HCl (Confab Laboratories) fasting (Experimental)
  Interventions: Drug: Tramadol hydrochloride
- 2: Tramadol HCl (Confab Laboratories) fed (Experimental)
  Interventions: Drug: Tramadol HCl
- 3: Tramadol HCl (Trillium Healthcare) fasting (Experimental)
  Interventions: Drug: Tramadol HCl

INTERVENTIONS:
Drug: Tramadol hydrochloride — 1x300mg Tramadol Hydrochloride (HCl) tablet (Confab Laboratories), fasting condition. Taken for one treatment period only, then subjects switched treatment at each period as per randomization schedule. Results are presented per treatment group overall.
  Arms: 1: Tramadol HCl (Confab Laboratories) fasting
Drug: Tramadol HCl — 1x300mg Tramadol Hydrochloride (HCl) tablet (Confab Laboratories), fed condition. Taken for one treatment period only, then subjects switched treatment at each period as per randomization schedule. Results are presented per treatment group overall.
  Arms: 2: Tramadol HCl (Confab Laboratories) fed
Drug: Tramadol HCl — 1x300mg Tramadol Hydrochloride (HCl) tablet (Trillium Healthcare) fasting condition. Taken for one treatment period only, then subjects switched treatment at each period as per randomization schedule. Results are presented per treatment group overall.
  Arms: 3: Tramadol HCl (Trillium Healthcare) fasting

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of two Tramadol Contramid® OAD 300 mg controlled-release tablets from two different manufacturing sites, administered as 1 x 300 mg controlled-release tablet under fasting conditions. The effect of food on the to-be-marketed formulation was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, non-smoker, ≥18 and ≤55 years of age.
* Capable of consent.
* Body Mass Index (BMI) ≥19.0 and <30.0 kg/m2.

Exclusion Criteria:

* Clinically significant illness or surgery within 4 weeks prior to dosing.
* Any clinically significant abnormality or abnormal laboratory test results found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Positive test for hepatitis B, hepatitis C, or HIV at screening.
* Electrocardiogram (ECG) abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 beats per minute [bpm]) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to tramadol or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (Selective serotonin reuptake inhibitors [SSRIs]), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to dosing.
* Clinically significant history or presence of any gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption and hormonal contraceptives.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 3 months preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:
* 50 mL to 499 mL of whole blood within 30 days,
* more than 499 mL of whole blood within 56 days prior to drug administration.
* Consumption of food or beverages containing grapefruit (e.g. fresh, canned, or frozen) within 7 days prior to administration of the study medication.
* History or presence of substance addiction.
* History of anaphylactoid reactions to codeine and other opioids.
* History of respiratory depression.
* History of increased intracranial pressure or head injury.
* History or presence of asthma, chronic obstructive pulmonary disease or other pulmonary condition that may predispose to hypoventilation.
* Opioid consumption in the 3 months preceding drug administration or history of drug dependence to any opioids.
* Positive urine pregnancy test at screening.
* Breast-feeding subject.
* Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 days prior to study drug administration. Acceptable methods of contraception are:
* intra-uterine contraceptive device (placed at least 4 weeks prior to study drug administration;
* condom or diaphragm + spermicide;
* hormonal contraceptives (starting at least 4 weeks prior to study drug administration).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2006-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

REFERENCES:
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Groups:
- Confab Fasting / Confab Fed / Trillium Fasting: Confab fasting / Confab fed / Trillium fasting Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1 x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 1, 1x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 2, and 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 3.
- Confab Fasting / Trillium Fasting / Confab Fed: Confab fasting / Trillium fasting / Confab fed Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1 x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 1, 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 2, and 1x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 3.
- Confab Fed / Confab Fasting / Trillium Fasting: Confab fasting / Trillium fasting / Confab fed Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 1, 1 x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 2, 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 3.
- Confab Fed / Trillium Fasting / Confab Fasting: Confab fed / Trillium fasting / Confab fasting Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 1, 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 2, and 1 x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 3.
- Trillium Fasting / Confab Fasting / Confab Fed: Trillium fasting / Confab fasting / Confab fed Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 1, 1 x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 2, and 1x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 3.
- Trillium Fasting / Confab Fed / Confab Fasting: Trillium fasting / Confab fasting / Confab fed Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 1, 1 x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 2, and 1x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 3.
Period: Treatment Period 1
Arm/Group | Confab Fasting / Confab Fed / Trillium Fasting | Confab Fasting / Trillium Fasting / Confab Fed | Confab Fed / Confab Fasting / Trillium Fasting | Confab Fed / Trillium Fasting / Confab Fasting | Trillium Fasting / Confab Fasting / Confab Fed | Trillium Fasting / Confab Fed / Confab Fasting
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 5 (One subject completed all of treatment period 1 assessments but did not enter treatment period 2) | 6 | 5 (One subject completed all of treatment period 1 assessments but did not enter treatment period 2) | 6 | 6
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0
Period: Treatment Period 2
Arm/Group | Confab Fasting / Confab Fed / Trillium Fasting | Confab Fasting / Trillium Fasting / Confab Fed | Confab Fed / Confab Fasting / Trillium Fasting | Confab Fed / Trillium Fasting / Confab Fasting | Trillium Fasting / Confab Fasting / Confab Fed | Trillium Fasting / Confab Fed / Confab Fasting
Started | 6 | 5 | 6 | 5 | 6 | 6
Completed | 6 | 5 | 5 (One subject completed treatment period 2 but did not enter treatment period 3) | 5 | 5 (One subject completed treatment period 2 but did not enter treatment period 3) | 6
Not Completed | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1 | 0
Period: Treatment Period 3
Arm/Group | Confab Fasting / Confab Fed / Trillium Fasting | Confab Fasting / Trillium Fasting / Confab Fed | Confab Fed / Confab Fasting / Trillium Fasting | Confab Fed / Trillium Fasting / Confab Fasting | Trillium Fasting / Confab Fasting / Confab Fed | Trillium Fasting / Confab Fed / Confab Fasting
Started | 6 | 5 | 5 | 5 | 5 | 6
Completed | 6 | 5 | 5 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Confab Fed / Confab Fasting / Trillium Fasting: Confab fed / Confab fasting / Trillium fasting Group includes patients receiving once daily administration of the following Tramadol Hydrochloride (HCl) treatment: 1x 300 mg tablet manufactured at Confab Laboratories, fed condition in treatment period 1, 1 x 300 mg tablet manufactured at Confab Laboratories, fasting condition in treatment period 2, 1 x 300 mg tablet manufactured at Trillium Healthcare Inc., fasting condition in treatment period 3.
- Total: Total of all reporting groups
Arm/Group | Confab Fasting / Confab Fed / Trillium Fasting | Confab Fasting / Trillium Fasting / Confab Fed | Confab Fed / Confab Fasting / Trillium Fasting | Confab Fed / Trillium Fasting / Confab Fasting | Trillium Fasting / Confab Fasting / Confab Fed | Trillium Fasting / Confab Fed / Confab Fasting | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 4 | 2 | 4 | 21
  Male | 2 | 3 | 2 | 2 | 4 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: AUC(0-t)
Description: Area under the plasma concentration (AUC) versus time curve to the last measurable concentration.
Time Frame: 48 hours
Population: Data from all randomized subjects who completed at least 2 periods of the study are presented.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Groups:
- 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting: Tramadol HCl 300 mg (Confab Laboratories) fasting Group includes the treatment period 1 data from subjects in the Confab fasting / Confab fed / Trillium fasting and Confab fasting / Trillium fasting / Confab fed sequences at period 1, plus the treatment period 2 data from subjects in the Confab fed / Confab fasting / Trillium fasting and Trillium fasting / Confab fasting / Confab fed sequences at period 2, and plus the treatment period 3 data from subjects in the Confab fed / Trillium fasting / Confab fasting and Trillium fasting / Confab fed / Confab fasting sequences at period 3.
- 2: Tramadol HCl 300 mg (Confab Laboratories) Fed: Tramadol HCl 300 mg (Confab Laboratories) fed Group includes the treatment period 1 data from subjects in the Confab fed / Confab fasting / Trillium fasting and Confab fed / Trillium fasting / Confab fasting sequences at period 1, plus the treatment period 2 data from subjects in the Confab fasting / Confab fed / Trillium fasting and Trillium fasting / Confab fed / Confab fasting sequences at period 2, and plus the treatment period 3 data from subjects in the Confab fasting / Trillium fasting / Confab fed and Trillium fasting / Confab fasting / Confab fed sequences at period 3.
- 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting: Tramadol HCl 300 mg (Trillium Healthcare) fasting Group includes the treatment period 1 data from subjects in the Trillium fasting / Confab fasting / Confab fed and Trillium fasting / Confab fed / Confab fasting sequences at period 1, plus the treatment period 2 data from subjects in the Confab fasting / Trillium fasting / Confab fed and Confab fed / Trillium fasting / Confab fasting sequences at period 2, and plus the treatment period 3 data from subjects in the Confab fasting / Confab fed / Trillium fasting and Confab fed / Confab fasting / Trillium fasting sequences at period 3.
Arm/Group | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting
Number analyzed (Participants) | 34 | 33 | 33
ng.h/mL | 9708 (3875) | 9696 (3750) | 9431 (3225)

2. Primary Outcome: AUC(0-∞)
Description: The area under the plasma concentration (AUC) curve was estimated by extrapolating to infinity AUC0-t. The extrapolation to infinity was done by regression with the last log-transformed data to estimate the terminal area by means of the line that maximized R'2 (coefficient of determination). The units are ng.h/mL.
  h=hours
Time Frame: 48 hours
Population: Data from all randomized subjects who completed at least 2 periods of the study are presented. The pharmacokinetic variables AUC(0-∞) of one subject for Tramadol HCl 300 mg (Confab Laboratories) fasting were not used in the analyses due to the morphology of the plasma concentration-time curves.
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting
Number analyzed (Participants) | 33 | 33 | 33
ng.h/mL | 9882 (3933) | 9898 (3970) | 10095 (4070)

3. Primary Outcome: Cmax
Description: Maximum plasma concentration (Cmax)
Time Frame: 48 hours
Population: Data from all randomized subjects who completed at least 2 periods of the study are presented.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting
Number analyzed (Participants) | 34 | 33 | 33
ng/mL | 433 (206) | 728 (317) | 402 (201)

4. Secondary Outcome: Tmax
Description: Time to maximum plasma concentration (Tmax)
Time Frame: 48 hours
Population: Data from all randomized subjects who completed at least 2 periods of the study are presented.
Measure: Median (Full Range); unit: hours
Arm/Group | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting
Number analyzed (Participants) | 34 | 33 | 33
hours | 7 [2 to 24] | 8 [3 to 20] | 12 [3 to 24]

5. Secondary Outcome: t1/2
Description: Apparent terminal elimination half-life (t1/2)
Time Frame: 48 hours
Population: Data from all randomized subjects who completed at least 2 periods of the study are presented. The pharmacokinetic variable T1/2 of one subject for Tramadol HCl 300 mg (Confab Laboratories) fasting were not used in the analyses due to the morphology of the plasma concentration-time curves.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting
Number analyzed (Participants) | 33 | 33 | 33
hours | 7.70 (1.97) | 6.61 (1.66) | 8.32 (2.84)

ADVERSE EVENTS:
Arm/Group | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 27/36 | 27/36 | 19/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Tramadol HCl 300 mg (Confab Laboratories) Fasting (N=36) | 2: Tramadol HCl 300 mg (Confab Laboratories) Fed (N=36) | 3: Tramadol HCl 300 mg (Trillium Healthcare) Fasting (N=36)
Difficulty to concentrate (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Difficulty voiding bladder (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 12 (12) | 11 (13) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2)
Feels euphoric (Psychiatric disorders) | 4 (4) | 4 (4) | 2 (2)
Feels sleepy (Nervous system disorders) | 7 (7) | 7 (7) | 6 (6)
Headache (General disorders) | 3 (3) | 7 (7) | 3 (3)
Hot flashes (Cardiac disorders) | 3 (3) | 6 (6) | 5 (5)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 13 (14) | 9 (9)
Stomach ache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (8) | 10 (10) | 8 (8)
Weakness (General disorders) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the study results may only be allowed with written permission from the sponsor.